CLINICAL TRIAL: NCT06381674
Title: Wearable Technology to Characterize and Treat mTBI Subtypes: Biofeedback-Based Precision Rehabilitation
Acronym: SuBTyPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laurie King, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHSU: 25890; HT9425-23-1-0845 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-04-04; First posted 2024-04-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Mild Traumatic Brain Injury, Concussion; Rehabilitation; Balance Impairment
Keywords: mild traumatic brain injury (mTBI); concussion; vestibular; ocular; balance; rehabilitation; biofeedback; wearable sensors
MeSH Terms: conditions — Brain Concussion | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: There will be two groups in this study that will be randomized concurrently into two different rehabilitation programs.
Who Masked: Outcomes Assessor
Masking Description: Parties that will be masked include those collecting and analyzing data before and after rehabilitation (post-doctorate fellows, research assistants, and statistician).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vestibular Therapy Augmented with Audio and Visual Real-Time Biofeedback (Experimental): This arm will receive 12 sessions over 6-weeks of vestibular therapy for mTBI (concussion) based on clinical practice guidelines augmented with visual and audio real-time biofeedback.
  Interventions: Other: Vestibular therapy for mTBI augmented with audio and visual real-time biofeedback
- Vestibular Therapy-Standard of Care (Active Comparator): This arm will receive 12 sessions of vestibular physical therapy over 6-weeks based on clinical practice guidelines for mTBI (concussion).
  Interventions: Other: Vestibular therapy for mTBI

INTERVENTIONS:
Other: Vestibular therapy for mTBI augmented with audio and visual real-time biofeedback — During physical therapy sessions participants will wear sensors on their head, chest, waist, and feet for real-time instrumented audio and visual biofeedback on quality of therapeutic exercise.
  Other Names: Rehabilitation
  Arms: Vestibular Therapy Augmented with Audio and Visual Real-Time Biofeedback
Other: Vestibular therapy for mTBI — During physical therapy sessions participants will go through vestibular therapeutic exercise WITHOUT audio and visual real-time biofeedback.
  Other Names: Rehabilitation
  Arms: Vestibular Therapy-Standard of Care

SUMMARY:
Current clinical assessment tools are often not sensitive enough to detect and treat some subtle (yet troubling) problems after mTBI. In this study, the investigators will use wearable sensors to both assess and treat people with mTBI. Specifically, the investigators will provide immediate feedback, with visual and/or auditory, on movement quality during physical therapy. This immediate feedback on performance may improve outcomes as the investigators will measure multiple body segments including head movements simultaneously with balance and walking exercises. Such complex movements are needed for safe return to high level activity and military duty. The investigators will test this approach against a standard vestibular rehabilitation program. There are few potential risks to this study such as increasing symptoms and a small fall risk. Benefits include physical therapy for balance problems regardless of therapy with or without biofeedback. An indirect benefit is to have data on correct dosage of physical therapy. The investigators will also distinguish which concussion subtype profiles benefit most from physical therapy. This will help healthcare providers and patients by providing more information to help establish clinical guidelines and new tools for physical therapy.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI) is common and can cause long-term problems. Balance problems are one of the most common problems and can prevent people from returning to their previous quality of life. People with mTBI can have many symptoms that present differently (i.e., 'subtypes'), making it difficult to evaluate and treat. Subtypes include cognitive, ocular-motor (vision problems), headache, vestibular (balance and dizziness) and mood. Correct detection of subtypes is important for patients to get the best and most specific (to their subtype) care, as quickly as possible. Our group has expertise in the subtypes that could likely affect balance and gait (vestibular and ocular-motor; V/O) and investigators plan to use wearable sensors and objective measures to improve detection and treatment of the problems that commonly occur in these subtypes. The investigators will test an approach (multi-segmental biofeedback) using wearable sensors that can measure how people move overall and can provide immediate feedback on how multiple body segments move during vestibular rehabilitation. Specifically, these sensors can provide feedback on head and body movement and speed but also measure how stable balance and walking are during an exercise. The investigators believe real-time feedback during the exercises will improve the quality of rehabilitation, specifically for those patients with V/O subtypes. The investigators also want to explore whether people with V/O subtypes move differently in the real world. The investigators will do this by measuring daily life mobility over 7 days using wearable sensors.

The Aims of this project are:

1. Aim I. Multidimensional, real-time biofeedback for rehabilitation: To determine if multidimensional real-time biofeedback using novel wearable technology that measures head/trunk and balance/gait improves outcomes after rehabilitation compared to standard care. For this aim, the investigators will enroll 100 participants (50 from Oregon Health & Science University and 50 from University of Utah). People will be randomized into either vestibular physical therapy augmented with visual/audio real-time biofeedback or into vestibular therapy without real-time biofeedback. Participants will be tested before and after a 6-week (2x/week) rehabilitation program. Our primary outcome will be the Patient Global Impression of Change (PGIC). Secondary outcomes will include Subjective Patient-reported, Clinical Assessment, and Instrumented Assessment measures.
2. Responsiveness to rehabilitation; objective measures to identify V/O subtype. Aim II is a separate analysis based on the data collected in Aim I. For this Aim, the 100 participants from Aim 1 will be grouped according to severity of V/O symptoms. Here, the investigators will explore: a) the responsiveness to rehabilitation by level of V/O deficit and b) the strength of the relationship between Patient-reported and Clinical and Instrumented Assessments of V/O measures.
3. Daily life mobility in people with V/O subtype: To: a) determine if daily life mobility (quality of gait and turning) is impacted differently in people with high V/O deficits and b) calculate healthy normative data for daily life mobility measures in active duty military service members. For Aim III, 50 people from Aim I, divided equally with V/O HI and V/O LO, will wear instrumented socks (APDM Wearable Technologies) over 7 days. Daily life mobility (quantity and quality) will also be collected on 40 healthy active duty service members over 7 days at Fort Sam Houston (FSH) to facilitate next steps in using continuous monitoring as an outcome measure after mTBI in the military.

ELIGIBILITY:
Inclusion Criteria:

* For all Aims, participants may be either civilians, active duty military, or Veterans, and must:

  1. have a diagnosis of mTBI based on VA/DoD criteria
  2. be between 18-60 years old,
  3. be able to stand unassisted for 10 minutes at a time
  4. be outside of the acute stage (> 2 weeks post-concussion) but within 6 months of their most recent mTBI and still reporting symptoms
  5. have at least some measurable deficit in Vestibular/Ocular categories based on Concussion Profile Screen
  6. have sufficient vision (corrected or uncorrected) for unassisted reading and performance of everyday personal tasks and independent community ambulation
  7. have adequate hearing (without amplification) adequate for engaging in close-range personal or telephone conversation.

Exclusion Criteria:

* Participants must not:

  1. have had or currently have any other injury, medical, or neurological illness that could potentially explain balance or vision deficits (e.g., CNS disease, stroke, epilepsy, greater than mild TBI, Meniere's, bilateral vestibular loss, recent lower extremity or spine orthopedic injury that impairs mobility) this includes unresolved symptoms from previous concussions
  2. meet criteria for moderate to severe substance-use disorder within the past month, as defined by DSM-V
  3. display behavior that would significantly interfere with the validity of data collection or safety during the study
  4. be in significant pain during the evaluation (> 7/10 by patient subjective report)
  5. be a pregnant female (balance considerations)
  6. been hospitalized for any brain injuries (separate from the emergency department)
  7. have significant joint pain or recent musculoskeletal injury that limits walking or mobility
  8. have had any major surgeries in the past year or amputation
  9. use an assistive device
  10. unable to stand barefoot
  11. currently receiving rehabilitation services for their mTBI or injuries related to their concussion (if rehabilitation has been completed more than 1 month ago participants may still be included).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) | Week 8 of study
  This single questionnaire will ask the participant to rate how they perceive their health has changed over the course of treatment. This scale is 1-7 where 1 is no change in quality of life and 7 is a great change that has made all the difference.

SECONDARY OUTCOMES:
Concussion Clinical Profiles Screening (CP Screening) | Weeks 1 and 8 of study
  This is a 29-item scale that is organized around concussion clinical profiles: 1) anxiety/mood (5 items), 2) cognitive/fatigue (3 items), 3) migraine (5 items), 4) ocular (5 items), and 5) vestibular (5 items); and 2 modifiers: 1) sleep (4 items), and 2) neck (cervical) (2 items). Participants respond to each item on a 0 (none) to 3 (severe) Likert-type scale. The CP Screen provides a total symptom score ranging from 0 to 87 and individual subscale scores. A higher score indicates a higher severity of symptoms.
Dizziness Handicap Index (DHI) | Weeks 1 and 8 of study
  This is a 25-item self-assessment inventory that evaluates the self-perceived handicapping effects due to a vestibular disorder. For scoring, 16-34 points is mild handicap, 36-52 points is a moderate handicap, and 54+ points severe handicap.
Quality of Life After Brain Injury (QOLIBRI) | Weeks 1 and 8 of study
  This is a questionnaire with 37 items addressing 6 dimensions of quality of life; cognition, self, daily life and autonomy, social relationships, physical problems and feeling bothered by emotions.The questionnaire provides a profile of quality of life together with a total score. It is easy to fill in, and can be completed in 7-10 minutes. The scale means are converted to the 0-100 scale by subtracting 1 from the mean and then multiplying by 25. This produces scale scores which have a lowest possible value of 0 (worst possible quality of life) and a maximum value of 100 (best possible quality of life).
The Patient Reported Outcomes Measurement Information System (PROMIS)-Satisfaction with Participation in Social Roles-Short Form 4a | Weeks 1 and 8 of study
  This is a questionnaire related to how satisfied participants are with social roles in the past 7 days. Higher scores mean more of the concept being measured. Example = more satisfaction.
Hospital Anxiety and Depression Scale (HADS) | Weeks 1 and 8 of study
  The HADS delineates potential anxiety or depression dominance where possible scores could range from 0 to 21 for anxiety and 0 to 21 for depression. Anxiety and depression are scored separately (8-10= mild, 11-14= moderate, 15-21= severe).
Headache Impact Test (HIT-6) | Weeks 1 and 8 of study
  This is a questionnaire that assesses the impact of headache severity on daily life activities. Higher scores indicate a greater impact on in the participant's life and the score range is 36-78. For example, a score of 36 is no impact on the participant's life and a score of 78 is always impacting the participant's life.
Insomnia Severity Index (ISI) | Weeks 1 and 8 of study
  This is 7-question survey that assess sleep problems. Respondents rate each element of the questionnaire using Likert-type scales. Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. Scores are tallied and can be compared both to scores obtained at a different phase of treatment and to the scores of other individuals. Though developers point out that their chosen cutoff scores have not been validated, they offer a few guidelines for interpreting scale results: a total score of 0-7 indicates no clinically significant insomnia, 8-14 means subthreshold insomnia, 15-21 is clinical insomnia (moderate severity), and 22-28 means clinical insomnia (severe).
Neck Disability Index (NDI) | Weeks 1 and 8 of study
  This questionnaire has 10 questions regarding neck pain during daily activities. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst. Alternately, the score can be reported from 0-100. The score is often reported as a percentage (0-100%).
Convergence Insufficiency Symptom Survey (CISS) | Weeks 1 and 8 of study
  This survey has 15 questions related to problems with convergence in everyday activities. Participants rate their symptoms on a 0-4 Likert Scale were 0 is never and 4 is always. A score of 21 or higher is suggestive of convergence insufficiency.
Vertigo Symptom Scale (VSS) | Weeks 1 and 8 of study
  The VSS contains 36 items addressing the frequency and severity of dizziness symptoms within the last 12 months. Frequency of symptoms is rated on a Likert scale: 0 points: "never", 1 point: "a few times (1-3 times a year)", 2 points: "several times (4-12 times a year)", 3 points: "quite often (on average, more than once a month)" and 4 points: "very often (on average more than once a week)". Total score aims to figure out the severity of dizziness where lower scores imply less severity. Two principle subscales are distinguishing between items related to vertigo and imbalance (Vertigo symptom scale) and those suggestive of anxiety and arousal (Autonomic/Anxiety).
  Vertigo/balance sub scale score range: 0-76 Autonomic/Anxiety subscale score range: 0-60
Automated Neuropsychological Assessment Metric (ANAM) | Weeks 1 and 8 of study
  This is a computerized neurocognitive test that takes about 20 minutes to complete. The ANAM collects information on attention, memory, or thinking ability.
Dynamic Visual Acuity ( DVA-Clinical) | Weeks 1 and 8 of study
  This test assesses gaze stability during head rotations relative to head-stationary visual acuity. The change in lines read compared to static acuity is noted. A loss of three or more lines of visual acuity relative to one's static visual acuity is regarded as clinically significant.
Ocular Motor Function Tests | Weeks 1 and 8 of study
  These tests will ask the participant to move their eyes in various directions.
Video Head Impulse Test (vHIT) | Weeks 1 and 8 of study
  This test will have the participant looking at a stationary object while their head is moved quickly.
Functional Gait Assessment (FGA) | Weeks 1 and 8 of study
  This assessment evaluates a patient's ability to adapt their balance while walking and undertaking a series of additional tasks such as turning their head, changing speeds, and stepping over an obstacle. Each item is scored on an ordinal scale from 0 to 3, with 0 = severe impairment, 1 = moderate impairment, 2 = mild impairment, 3 = normal ambulation and highest score = 30.
Complex Turning Course (CTC) | Weeks 1 and 8 of study
  This is a test of mobility that evaluates a person's ability to walk a prescribed path involving multiple turns of various angles.
Modified Balance Error Scoring System (mBESS) | Weeks 1 and 8 of study
  This test assesses balance by asking participants to stand in progressively challenging conditions (feet together, single limb stance and tandem) both on firm and foam surfaces. All items are performed with eyes closed. A rater evaluates the number of errors committed by the participant, such as opening their eyes or removing their hands from their hips during the first 20 seconds of the trial for each test. The total score can be between 0-30, where a higher score indicates more errors.
Modified Clinical Test for Sensory Integration on Balance (mCTSIB) | Weeks 1 and 8 of study
  This test assesses the sensory contributions to balance. In this test, participants stand with feet together in 4 conditions; 1) eyes open on a firm surface, 2) eyes closed on a firm surface, 3) eyes open on foam surface, and 4) eyes closed on a foam surface. Participants are clinician-rated on stability based on the ability to maintain balance for 30 seconds in each condition. If the subject cannot hold the position the test is stopped and the time is recorded for each trial. Completing 30 seconds for each trial is the optimal score. Total time is recorded, 120 seconds is optimal.
Instrumented One Minute Walk (Single and Dual Task) | Weeks 1 and 8 of study
  This is a measurement of over-ground walking performance over 1 minute with and without additional cognitive tasks.
Hybrid Assessment of Mobility (HAM-4) | Weeks 1 and 8 of study
  This test includes two components of the FGA (horizontal head turns and gait with pivot turn), as well as a fast walk forward and backward from the HiMAT. The highest possible score is 14. The higher the score, the higher the level of performance.
Tandem Gait (Single and Dual Task) | Weeks 1 and 8 of study
  This test will ask the participant to perform heel-to-toe walking without separating heel and toe as accurately and quickly as they can with and without additional cognitive tasks. Participants must complete the task without separating heel and toe or other deviations. Time will be recorded of the passing trials. A lower time indicates better performance.
Vestibular Ocular Motor Screening (VOMS) | Weeks 1 and 8 of study
  This test will look at a patient's symptom provocation with various head and eye movements. Baseline symptoms will be assessed 0-10 where 0 is no symptoms and 10 is the maximum severity of symptoms. After each test the subject will be asked to rate their symptoms 0-10. Total Score and change scores are calculated where high scores indicate more severe symptoms.
Central Sensorimotor Integration Testing (CSMI) | Weeks 1 and 8 of study
  The participant will be tested on a modified Research NeuroCom platform where they will stand on a force plate to record postural sway. The surface and/or visual surround will move while they will be instructed to maintain their balance. They will wear a safety harness attached above to prevent falling in case a loss of balance occurs.
Reactive Balance | Weeks 1 and 8 of study
  The participant will be tested on their reactive stepping in the anterior, posterior, and lateral directions.
Neurobehavioral Symptoms Inventory (NSI) | Weeks 1 and 8 of the study.
  This questionnaire has 22 questions and asks participants to rate how much a symptom disturbed them from 0 (none) to 3 (severe) over the past two weeks. The total score is the sum of responses.
International Physical Activity Questionnaire (IPAQ) | Weeks 1 and 8 of study.
  This questionnaire assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A King, PhD, DPT, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Oregon Health & Science University, Portland, Oregon
  - Fort Sam Houston, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] The Management and Rehabilitation of Post-Acute Mild Traumatic Brain Injury Work Group. VA/DoD Clinical Practice Guidelines for the Management of Concussion-Mild Traumatic Brain Injury. 2021:1-128.
- [Background] Silverberg ND, Iaccarino MA, Panenka WJ, Iverson GL, McCulloch KL, Dams-O'Connor K, Reed N, McCrea M; American Congress of Rehabilitation Medicine Brain Injury Interdisciplinary Special Interest Group Mild TBI Task Force. Management of Concussion and Mild Traumatic Brain Injury: A Synthesis of Practice Guidelines. Arch Phys Med Rehabil. 2020 Feb;101(2):382-393. doi: 10.1016/j.apmr.2019.10.179. Epub 2019 Oct 23. PMID 31654620
- [Background] Coronado VG, McGuire LC, Sarmiento K, Bell J, Lionbarger MR, Jones CD, Geller AI, Khoury N, Xu L. Trends in Traumatic Brain Injury in the U.S. and the public health response: 1995-2009. J Safety Res. 2012 Sep;43(4):299-307. doi: 10.1016/j.jsr.2012.08.011. Epub 2012 Aug 25. PMID 23127680
- [Background] Corso P, Finkelstein E, Miller T, Fiebelkorn I, Zaloshnja E. Incidence and lifetime costs of injuries in the United States. Inj Prev. 2006 Aug;12(4):212-8. doi: 10.1136/ip.2005.010983. PMID 16887941
- [Background] Vanderploeg RD, Curtiss G, Luis CA, Salazar AM. Long-term morbidities following self-reported mild traumatic brain injury. J Clin Exp Neuropsychol. 2007 Aug;29(6):585-98. doi: 10.1080/13803390600826587. PMID 17691031
- [Background] Walker WC, Nowak KJ, Kenney K, Franke LM, Eapen BC, Skop K, Levin H, Agyemang AA, Tate DF, Wilde EA, Hinds S, Nolen TL. Is balance performance reduced after mild traumatic brain injury?: Interim analysis from chronic effects of neurotrauma consortium (CENC) multi-centre study. Brain Inj. 2018;32(10):1156-1168. doi: 10.1080/02699052.2018.1483529. Epub 2018 Jun 12. PMID 29894203
- [Background] McCrory P. Sports concussion and the risk of chronic neurological impairment. Clin J Sport Med. 2011 Jan;21(1):6-12. doi: 10.1097/JSM.0b013e318204db50. PMID 21200164
- [Background] Guskiewicz KM, McCrea M, Marshall SW, Cantu RC, Randolph C, Barr W, Onate JA, Kelly JP. Cumulative effects associated with recurrent concussion in collegiate football players: the NCAA Concussion Study. JAMA. 2003 Nov 19;290(19):2549-55. doi: 10.1001/jama.290.19.2549. PMID 14625331
- [Background] Kardouni JR, Shing TL, McKinnon CJ, Scofield DE, Proctor SP. Risk for Lower Extremity Injury After Concussion: A Matched Cohort Study in Soldiers. J Orthop Sports Phys Ther. 2018 Jul;48(7):533-540. doi: 10.2519/jospt.2018.8053. Epub 2018 May 8. PMID 29739302
- [Background] Fino PC, Becker LN, Fino NF, Griesemer B, Goforth M, Brolinson PG. Effects of Recent Concussion and Injury History on Instantaneous Relative Risk of Lower Extremity Injury in Division I Collegiate Athletes. Clin J Sport Med. 2019 May;29(3):218-223. doi: 10.1097/JSM.0000000000000502. PMID 31033615
- [Background] McPherson AL, Nagai T, Webster KE, Hewett TE. Musculoskeletal Injury Risk After Sport-Related Concussion: A Systematic Review and Meta-analysis. Am J Sports Med. 2019 Jun;47(7):1754-1762. doi: 10.1177/0363546518785901. Epub 2018 Aug 3. PMID 30074832
- [Background] Murray DA, Meldrum D, Lennon O. Can vestibular rehabilitation exercises help patients with concussion? A systematic review of efficacy, prescription and progression patterns. Br J Sports Med. 2017 Mar;51(5):442-451. doi: 10.1136/bjsports-2016-096081. Epub 2016 Sep 21. PMID 27655831
- [Background] Carter KM, Pauhl AN, Christie AD. The Role of Active Rehabilitation in Concussion Management: A Systematic Review and Meta-analysis. Med Sci Sports Exerc. 2021 Sep 1;53(9):1835-1845. doi: 10.1249/MSS.0000000000002663. PMID 33787531
- [Background] Reid SA, Farbenblum J, McLeod S. Do physical interventions improve outcomes following concussion: a systematic review and meta-analysis? Br J Sports Med. 2022 Mar;56(5):292-298. doi: 10.1136/bjsports-2020-103470. Epub 2021 Sep 30. PMID 34593371
- [Background] Paul SS, Dibble LE, Walther RG, Shelton C, Gurgel RK, Lester ME. Characterization of Head-Trunk Coordination Deficits After Unilateral Vestibular Hypofunction Using Wearable Sensors. JAMA Otolaryngol Head Neck Surg. 2017 Oct 1;143(10):1008-1014. doi: 10.1001/jamaoto.2017.1443. PMID 28859201
- [Background] Paul SS, Dibble LE, Walther RG, Shelton C, Gurgel RK, Lester ME. Reduced Purposeful Head Movements During Community Ambulation Following Unilateral Vestibular Loss. Neurorehabil Neural Repair. 2018 Apr-May;32(4-5):309-316. doi: 10.1177/1545968318770271. Epub 2018 Apr 20. PMID 29676210
- [Background] Fino PC, Wilhelm J, Parrington L, Stuart S, Chesnutt JC, King LA. Inertial Sensors Reveal Subtle Motor Deficits When Walking With Horizontal Head Turns After Concussion. J Head Trauma Rehabil. 2019 Mar/Apr;34(2):E74-E81. doi: 10.1097/HTR.0000000000000418. PMID 30045224
- [Background] Konrad HR, Tomlinson D, Stockwell CW, Norre M, Horak FB, Shepard NT, Herdman SJ. Rehabilitation therapy for patients with disequilibrium and balance disorders. Otolaryngol Head Neck Surg. 1992 Jul;107(1):105-8. doi: 10.1177/019459989210700117. PMID 1528589
- [Background] Cabrera Kang CM, Tusa RJ. Vestibular rehabilitation: rationale and indications. Semin Neurol. 2013 Jul;33(3):276-85. doi: 10.1055/s-0033-1354593. Epub 2013 Sep 21. PMID 24057831
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496
- [Background] Loyd BJ, Saviers-Steiger J, Fangman A, Ballard P, Taylor C, Schubert M, Dibble L. Turning Toward Monitoring of Gaze Stability Exercises: The Utility of Wearable Sensors. J Neurol Phys Ther. 2020 Oct;44(4):261-267. doi: 10.1097/NPT.0000000000000329. PMID 32815892
- [Background] Martini DNP, Wilhelm, J.L., Parrington, L., King, L.A. Wearable Sensors for Vestibular Rehabilitation: A Pilot Study. Journal of Physiotherapy Research. 2021; 5(8):31.
- [Background] Winstein CJ. Knowledge of results and motor learning--implications for physical therapy. Phys Ther. 1991 Feb;71(2):140-9. doi: 10.1093/ptj/71.2.140. PMID 1989009
- [Background] Zhou Y, Shao W, Wang L. Effects of Feedback on Students' Motor Skill Learning in Physical Education: A Systematic Review. Int J Environ Res Public Health. 2021 Jun 10;18(12):6281. doi: 10.3390/ijerph18126281. PMID 34200657
- [Background] Adams JA. A closed-loop theory of motor learning. J Mot Behav. 1971 Jun;3(2):111-49. doi: 10.1080/00222895.1971.10734898. PMID 15155169
- [Background] Dozza M, Chiari L, Horak FB. Audio-biofeedback improves balance in patients with bilateral vestibular loss. Arch Phys Med Rehabil. 2005 Jul;86(7):1401-3. doi: 10.1016/j.apmr.2004.12.036. PMID 16003671
- [Background] Moore S, Woollacott M. The use of biofeedback devices to improve postural stability. Phys Ther Pract. 1993;2(2):1-19.
- [Background] Bowman T, Gervasoni E, Arienti C, Lazzarini SG, Negrini S, Crea S, Cattaneo D, Carrozza MC. Wearable Devices for Biofeedback Rehabilitation: A Systematic Review and Meta-Analysis to Design Application Rules and Estimate the Effectiveness on Balance and Gait Outcomes in Neurological Diseases. Sensors (Basel). 2021 May 15;21(10):3444. doi: 10.3390/s21103444. PMID 34063355
- [Background] Hebert JR, Forster JE, Stearns-Yoder KA, Penzenik ME, Brenner LA. Persistent Symptoms and Objectively Measured Balance Performance Among OEF/OIF Veterans With Remote Mild Traumatic Brain Injury. J Head Trauma Rehabil. 2018 Nov/Dec;33(6):403-411. doi: 10.1097/HTR.0000000000000385. PMID 29385020
- [Background] Herdman SJ, Tusa RJ, Blatt P, Suzuki A, Venuto PJ, Roberts D. Computerized dynamic visual acuity test in the assessment of vestibular deficits. Am J Otol. 1998 Nov;19(6):790-6. PMID 9831156
- [Background] Quintana C, Heebner NR, Olson AD, Abt JP, Hoch MC. Sport-specific differences in dynamic visual acuity and gaze stabilization in division-I collegiate athletes. J Vestib Res. 2020;30(4):249-257. doi: 10.3233/VES-200710. PMID 32925127
- [Background] Collins MW, Kontos AP, Reynolds E, Murawski CD, Fu FH. A comprehensive, targeted approach to the clinical care of athletes following sport-related concussion. Knee Surg Sports Traumatol Arthrosc. 2014 Feb;22(2):235-46. doi: 10.1007/s00167-013-2791-6. Epub 2013 Dec 12. PMID 24337463
- [Background] Kontos A. Concussion: A clinical profile approach to assessment and treatment. New Ed: American Psychological Association; 2018.
- [Background] Langdon S, Konigs M, Adang EAMC, Goedhart E, Oosterlaan J. Subtypes of Sport-Related Concussion: a Systematic Review and Meta-cluster Analysis. Sports Med. 2020 Oct;50(10):1829-1842. doi: 10.1007/s40279-020-01321-9. PMID 32720230
- [Background] Lumba-Brown A, Teramoto M, Bloom OJ, Brody D, Chesnutt J, Clugston JR, Collins M, Gioia G, Kontos A, Lal A, Sills A, Ghajar J. Concussion Guidelines Step 2: Evidence for Subtype Classification. Neurosurgery. 2020 Jan 1;86(1):2-13. doi: 10.1093/neuros/nyz332. PMID 31432081
- [Background] Kontos AP, Elbin RJ, Trbovich A, Womble M, Said A, Sumrok VF, French J, Kegel N, Puskar A, Sherry N, Holland C, Collins M. Concussion Clinical Profiles Screening (CP Screen) Tool: Preliminary Evidence to Inform a Multidisciplinary Approach. Neurosurgery. 2020 Aug 1;87(2):348-356. doi: 10.1093/neuros/nyz545. PMID 31950187
- [Background] Gioia G. Defining concussion subtype treatment targets: psychometric properties of the concussion symptom subtypes inventory (CSSI). International Child Neurology Association-CNS; San Diego, CA.2020.
- [Background] Lumba-Brown A, Ghajar J, Cornwell J, Bloom OJ, Chesnutt J, Clugston JR, Kolluri R, Leddy JJ, Teramoto M, Gioia G. Representation of concussion subtypes in common postconcussion symptom-rating scales. Concussion. 2019 Nov 1;4(3):CNC65. doi: 10.2217/cnc-2019-0005. PMID 31827883
- [Background] Riemann BL, Guskiewicz KM. Effects of mild head injury on postural stability as measured through clinical balance testing. J Athl Train. 2000 Jan;35(1):19-25. PMID 16558603
- [Background] Giza CC, Kutcher JS, Ashwal S, Barth J, Getchius TS, Gioia GA, Gronseth GS, Guskiewicz K, Mandel S, Manley G, McKeag DB, Thurman DJ, Zafonte R. Summary of evidence-based guideline update: evaluation and management of concussion in sports [RETIRED]: report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2013 Jun 11;80(24):2250-7. doi: 10.1212/WNL.0b013e31828d57dd. Epub 2013 Mar 18. PMID 23508730
- [Background] Finnoff JT, Peterson VJ, Hollman JH, Smith J. Intrarater and interrater reliability of the Balance Error Scoring System (BESS). PM R. 2009 Jan;1(1):50-4. doi: 10.1016/j.pmrj.2008.06.002. Epub 2008 Dec 10. PMID 19627872
- [Background] King LA, Horak FB, Mancini M, Pierce D, Priest KC, Chesnutt J, Sullivan P, Chapman JC. Instrumenting the balance error scoring system for use with patients reporting persistent balance problems after mild traumatic brain injury. Arch Phys Med Rehabil. 2014 Feb;95(2):353-9. doi: 10.1016/j.apmr.2013.10.015. Epub 2013 Nov 5. PMID 24200875
- [Background] Gera G, Chesnutt J, Mancini M, Horak FB, King LA. Inertial Sensor-Based Assessment of Central Sensory Integration for Balance After Mild Traumatic Brain Injury. Mil Med. 2018 Mar 1;183(suppl_1):327-332. doi: 10.1093/milmed/usx162. PMID 29635623
- [Background] Hasegawa N, Shah VV, Harker G, Carlson-Kuhta P, Nutt JG, Lapidus JA, Jung SH, Barlow N, King LA, Horak FB, Mancini M. Responsiveness of Objective vs. Clinical Balance Domain Outcomes for Exercise Intervention in Parkinson's Disease. Front Neurol. 2020 Sep 25;11:940. doi: 10.3389/fneur.2020.00940. eCollection 2020. PMID 33101161
- [Background] El-Gohary M, Pearson S, McNames J, Mancini M, Horak F, Mellone S, Chiari L. Continuous monitoring of turning in patients with movement disability. Sensors (Basel). 2013 Dec 27;14(1):356-69. doi: 10.3390/s140100356. PMID 24379043
- [Background] Mancini M, King L, Salarian A, Holmstrom L, McNames J, Horak FB. Mobility Lab to Assess Balance and Gait with Synchronized Body-worn Sensors. J Bioeng Biomed Sci. 2011 Dec 12;Suppl 1:007. doi: 10.4172/2155-9538.S1-007. PMID 24955286
- [Background] Shah VV, McNames J, Mancini M, Carlson-Kuhta P, Spain RI, Nutt JG, El-Gohary M, Curtze C, Horak FB. Quantity and quality of gait and turning in people with multiple sclerosis, Parkinson's disease and matched controls during daily living. J Neurol. 2020 Apr;267(4):1188-1196. doi: 10.1007/s00415-020-09696-5. Epub 2020 Jan 11. PMID 31927614
- [Background] Stuart S, Parrington L, Martini DN, Kreter N, Chesnutt JC, Fino PC, King LA. Analysis of Free-Living Mobility in People with Mild Traumatic Brain Injury and Healthy Controls: Quality over Quantity. J Neurotrauma. 2020 Jan 1;37(1):139-145. doi: 10.1089/neu.2019.6450. Epub 2019 Aug 26. PMID 31354032
- [Background] Brooke J. SUS: A Quick and Dirty Usability Scale. Usability Evaluation in Industry. 1996. CRC Press
- [Background] Brooke J. SUS: a retrospective. Journal of Usability Studies. 2013;8:29-40. 51.
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Powell D, Godfrey A, Parrington L, Campbell KR, King LA, Stuart S. Free-living gait does not differentiate chronic mTBI patients compared to healthy controls. J Neuroeng Rehabil. 2022 May 26;19(1):49. doi: 10.1186/s12984-022-01030-6. PMID 35619112
- [Background] Centers for Disease Control and Prevention. Report to congress on traumatic brain injury in the United States: epidemiology and rehabilitation. Atlanta, GA: National Center for Injury Prevention and Control; 2014.
- [Background] Assistant Secretary of Defense. Traumatic brain injury: Updated definition and reporting. Washington DC, Department of Defense; 2015.
- [Background] Hoffer ME, Gottshall K, Viirre ES. Vestibular Consequences of mTBI. in: traumatic brain injury: a clinician's guide to diagnosis, management, and rehabilitation. New York: Springer New York; 2012.139-47.
- [Background] Software NS. Power Analysis & Sample Size (PASS) 2019.
- [Background] Quatman-Yates CC, Hunter-Giordano A, Shimamura KK, Landel R, Alsalaheen BA, Hanke TA, McCulloch KL. Physical Therapy Evaluation and Treatment After Concussion/Mild Traumatic Brain Injury. J Orthop Sports Phys Ther. 2020 Apr;50(4):CPG1-CPG73. doi: 10.2519/jospt.2020.0301. PMID 32241234
- [Background] Jull G, Trott P, Potter H, Zito G, Niere K, Shirley D, Emberson J, Marschner I, Richardson C. A randomized controlled trial of exercise and manipulative therapy for cervicogenic headache. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1835-43; discussion 1843. doi: 10.1097/00007632-200209010-00004. PMID 12221344
- [Background] Leddy JJ, Kozlowski K, Donnelly JP, Pendergast DR, Epstein LH, Willer B. A preliminary study of subsymptom threshold exercise training for refractory post-concussion syndrome. Clin J Sport Med. 2010 Jan;20(1):21-7. doi: 10.1097/JSM.0b013e3181c6c22c. PMID 20051730
- [Background] Leddy JJ, Willer B. Use of graded exercise testing in concussion and return-to-activity management. Curr Sports Med Rep. 2013 Nov-Dec;12(6):370-6. doi: 10.1249/JSR.0000000000000008. PMID 24225521
- [Background] Grinnon ST, Miller K, Marler JR, Lu Y, Stout A, Odenkirchen J, Kunitz S. National Institute of Neurological Disorders and Stroke Common Data Element Project - approach and methods. Clin Trials. 2012 Jun;9(3):322-9. doi: 10.1177/1740774512438980. Epub 2012 Feb 27. PMID 22371630
- [Background] Kontos AP, Deitrick JM, Collins MW, Mucha A. Review of Vestibular and Oculomotor Screening and Concussion Rehabilitation. J Athl Train. 2017 Mar;52(3):256-261. doi: 10.4085/1062-6050-51.11.05. PMID 28387548
- [Background] Wilde EA, Whiteneck GG, Bogner J, Bushnik T, Cifu DX, Dikmen S, French L, Giacino JT, Hart T, Malec JF, Millis SR, Novack TA, Sherer M, Tulsky DS, Vanderploeg RD, von Steinbuechel N. Recommendations for the use of common outcome measures in traumatic brain injury research. Arch Phys Med Rehabil. 2010 Nov;91(11):1650-1660.e17. doi: 10.1016/j.apmr.2010.06.033. PMID 21044708
- [Background] Broglio SP, Kontos AP, Levin H, Schneider K, Wilde EA, Cantu RC, Feddermann-Demont N, Fuller GW, Gagnon I, Gioia GA, Giza C, Griesbach GS, Leddy JJ, Lipton ML, Mayer AR, McAllister TW, McCrea M, McKenzie LB, Putukian M, Signoretti S, Suskauer SJ, Tamburro R, Turner M, Yeates KO, Zemek R, Ala'i S, Esterlitz J, Gay K, Bellgowan PSF, Joseph K. National Institute of Neurological Disorders and Stroke and Department of Defense Sport-Related Concussion Common Data Elements Version 1.0 Recommendations. J Neurotrauma. 2018 Dec 1;35(23):2776-2783. doi: 10.1089/neu.2018.5643. Epub 2018 Jul 23. PMID 29717643
- [Background] Morris R, Stuart S, McBarron G, Fino PC, Mancini M, Curtze C. Validity of Mobility Lab (version 2) for gait assessment in young adults, older adults and Parkinson's disease. Physiol Meas. 2019 Sep 30;40(9):095003. doi: 10.1088/1361-6579/ab4023. PMID 31470423
- [Background] Tate DF, Dennis EL, Adams JT, Adamson MM, Belanger HG, Bigler ED, Bouchard HC, Clark AL, Delano-Wood LM, Disner SG, Eapen BC, Franz CE, Geuze E, Goodrich-Hunsaker NJ, Han K, Hayes JP, Hinds SR 2nd, Hodges CB, Hovenden ES, Irimia A, Kenney K, Koerte IK, Kremen WS, Levin HS, Lindsey HM, Morey RA, Newsome MR, Ollinger J, Pugh MJ, Scheibel RS, Shenton ME, Sullivan DR, Taylor BA, Troyanskaya M, Velez C, Wade BS, Wang X, Ware AL, Zafonte R, Thompson PM, Wilde EA. Coordinating Global Multi-Site Studies of Military-Relevant Traumatic Brain Injury: Opportunities, Challenges, and Harmonization Guidelines. Brain Imaging Behav. 2021 Apr;15(2):585-613. doi: 10.1007/s11682-020-00423-2. Epub 2021 Jan 7. PMID 33409819
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Gottshall K, Drake A, Gray N, McDonald E, Hoffer ME. Objective vestibular tests as outcome measures in head injury patients. Laryngoscope. 2003 Oct;113(10):1746-50. doi: 10.1097/00005537-200310000-00016. PMID 14520100
- [Background] Kaufman KR, Brey RH, Chou LS, Rabatin A, Brown AW, Basford JR. Comparison of subjective and objective measurements of balance disorders following traumatic brain injury. Med Eng Phys. 2006 Apr;28(3):234-9. doi: 10.1016/j.medengphy.2005.05.005. Epub 2005 Jul 25. PMID 16043377
- [Background] Basford JR, Chou LS, Kaufman KR, Brey RH, Walker A, Malec JF, Moessner AM, Brown AW. An assessment of gait and balance deficits after traumatic brain injury. Arch Phys Med Rehabil. 2003 Mar;84(3):343-9. doi: 10.1053/apmr.2003.50034. PMID 12638101
- [Background] Lin LF, Liou TH, Hu CJ, Ma HP, Ou JC, Chiang YH, Chiu WT, Tsai SH, Chu WC. Balance function and sensory integration after mild traumatic brain injury. Brain Inj. 2015;29(1):41-6. doi: 10.3109/02699052.2014.955881. PMID 25265292
- [Background] King PR, Donnelly KT, Donnelly JP, Dunnam M, Warner G, Kittleson CJ, Bradshaw CB, Alt M, Meier ST. Psychometric study of the Neurobehavioral Symptom Inventory. J Rehabil Res Dev. 2012;49(6):879-88. doi: 10.1682/jrrd.2011.03.0051. PMID 23299259
- [Background] von Steinbuchel N, Wilson L, Gibbons H, Hawthorne G, Hofer S, Schmidt S, Bullinger M, Maas A, Neugebauer E, Powell J, von Wild K, Zitnay G, Bakx W, Christensen AL, Koskinen S, Formisano R, Saarajuri J, Sasse N, Truelle JL; QOLIBRI Task Force. Quality of Life after Brain Injury (QOLIBRI): scale validity and correlates of quality of life. J Neurotrauma. 2010 Jul;27(7):1157-65. doi: 10.1089/neu.2009.1077. PMID 20210602
- [Background] Moore BM, Adams JT, Barakatt E. Outcomes Following a Vestibular Rehabilitation and Aerobic Training Program to Address Persistent Post-Concussion Symptoms. J Allied Health. 2016 Winter;45(4):e59-e68. PMID 27915363
- [Background] van der Naalt J, van Zomeren AH, Sluiter WJ, Minderhoud JM. One year outcome in mild to moderate head injury: the predictive value of acute injury characteristics related to complaints and return to work. J Neurol Neurosurg Psychiatry. 1999 Feb;66(2):207-13. doi: 10.1136/jnnp.66.2.207. PMID 10071101
- [Background] Shumway-Cook A, Horak FB. Assessing the influence of sensory interaction of balance. Suggestion from the field. Phys Ther. 1986 Oct;66(10):1548-50. doi: 10.1093/ptj/66.10.1548. No abstract available. PMID 3763708
- [Background] Pape MM, Kodosky PN, Hoover P. The Community Balance and Mobility Scale: Detecting Impairments in Military Service Members With Mild Traumatic Brain Injury. Mil Med. 2020 Mar 2;185(3-4):428-435. doi: 10.1093/milmed/usz265. PMID 31621858
- [Background] Pin TW. Psychometric properties of 2-minute walk test: a systematic review. Arch Phys Med Rehabil. 2014 Sep;95(9):1759-75. doi: 10.1016/j.apmr.2014.03.034. Epub 2014 May 9. PMID 24814460
- [Background] Fino PC, Weightman MM, Dibble LE, Lester ME, Hoppes CW, Parrington L, Arango J, Souvignier A, Roberts H, King LA. Objective Dual-Task Turning Measures for Return-to-Duty Assessment After Mild Traumatic Brain Injury: The ReTURN Study Protocol. Front Neurol. 2021 Jan 15;11:544812. doi: 10.3389/fneur.2020.544812. eCollection 2020. PMID 33519659
- [Background] Mucha A, Collins MW, Elbin RJ, Furman JM, Troutman-Enseki C, DeWolf RM, Marchetti G, Kontos AP. A Brief Vestibular/Ocular Motor Screening (VOMS) assessment to evaluate concussions: preliminary findings. Am J Sports Med. 2014 Oct;42(10):2479-86. doi: 10.1177/0363546514543775. Epub 2014 Aug 8. PMID 25106780
- [Background] Badke MB, Shea TA, Miedaner JA, Grove CR. Outcomes after rehabilitation for adults with balance dysfunction. Arch Phys Med Rehabil. 2004 Feb;85(2):227-33. doi: 10.1016/j.apmr.2003.06.006. PMID 14966706
- [Background] Dannenbaum E, Paquet N, Chilingaryan G, Fung J. Clinical evaluation of dynamic visual acuity in subjects with unilateral vestibular hypofunction. Otol Neurotol. 2009 Apr;30(3):368-72. doi: 10.1097/MAO.0b013e31819bda35. PMID 19318888
- [Background] Washabaugh EP, Kalyanaraman T, Adamczyk PG, Claflin ES, Krishnan C. Validity and repeatability of inertial measurement units for measuring gait parameters. Gait Posture. 2017 Jun;55:87-93. doi: 10.1016/j.gaitpost.2017.04.013. Epub 2017 Apr 12. PMID 28433867
- [Background] King LA, Mancini M, Fino PC, Chesnutt J, Swanson CW, Markwardt S, Chapman JC. Sensor-Based Balance Measures Outperform Modified Balance Error Scoring System in Identifying Acute Concussion. Ann Biomed Eng. 2017 Sep;45(9):2135-2145. doi: 10.1007/s10439-017-1856-y. Epub 2017 May 24. PMID 28540448
- [Background] Parrington L, King LA, Weightman MM, Hoppes CW, Lester ME, Dibble LE, Fino PC. Between-site equivalence of turning speed assessments using inertial measurement units. Gait Posture. 2021 Oct;90:245-251. doi: 10.1016/j.gaitpost.2021.09.164. Epub 2021 Sep 9. PMID 34530311
- [Background] Loyd BJ, Dibble LE, Weightman MM, Pelo R, Hoppes CW, Lester M, King LA, Fino PC. Volitional Head Movement Deficits and Alterations in Gait Speed Following Mild Traumatic Brain Injury. J Head Trauma Rehabil. 2023 May-Jun 01;38(3):E223-E232. doi: 10.1097/HTR.0000000000000831. Epub 2022 Oct 14. PMID 36731009
- [Background] Stuart S, Parrington L, Morris R, Martini DN, Fino PC, King LA. Gait measurement in chronic mild traumatic brain injury: A model approach. Hum Mov Sci. 2020 Feb;69:102557. doi: 10.1016/j.humov.2019.102557. Epub 2019 Nov 26. PMID 31783306
- [Background] Fino PC, Parrington L, Walls M, Sippel E, Hullar TE, Chesnutt JC, King LA. Abnormal Turning and Its Association with Self-Reported Symptoms in Chronic Mild Traumatic Brain Injury. J Neurotrauma. 2018 May 15;35(10):1167-1177. doi: 10.1089/neu.2017.5231. Epub 2018 Mar 23. PMID 29078732
- [Background] Blanchard EB, Jones-Alexander J, Buckley TC, Forneris CA. Psychometric properties of the PTSD Checklist (PCL). Behav Res Ther. 1996 Aug;34(8):669-73. doi: 10.1016/0005-7967(96)00033-2. PMID 8870294
- [Background] Ruggiero KJ, Del Ben K, Scotti JR, Rabalais AE. Psychometric properties of the PTSD Checklist-Civilian Version. J Trauma Stress. 2003 Oct;16(5):495-502. doi: 10.1023/A:1025714729117. PMID 14584634
- [Background] Kontos AP, Sufrinko A, Sandel N, Emami K, Collins MW. Sport-related Concussion Clinical Profiles: Clinical Characteristics, Targeted Treatments, and Preliminary Evidence. Curr Sports Med Rep. 2019 Mar;18(3):82-92. doi: 10.1249/JSR.0000000000000573. PMID 30855306
- [Background] Chan F, Gelman JS, Ditchman N, Kim J-H, Chiu C-Y. The World Health Organization ICF model as a conceptual framework of disability. Understanding psychosocial adjustment to chronic illness and disability: A handbook for evidence-based practitioners in rehabilitation. New York, NY, US: Springer Publishing Company; 2009. p. 23-50.
- [Background] Houston MN, Bay RC, Valovich McLeod TC. The relationship between post-injury measures of cognition, balance, symptom reports and health-related quality-of-life in adolescent athletes with concussion. Brain Inj. 2016;30(7):891-8. doi: 10.3109/02699052.2016.1146960. Epub 2016 Apr 18. PMID 27088297
- [Background] van Ierssel J, Sveistrup H, Marshall S. Identifying the concepts contained within health-related quality of life outcome measures in concussion research using the International Classification of Functioning, Disability, and Health as a reference: a systematic review. Qual Life Res. 2018 Dec;27(12):3071-3086. doi: 10.1007/s11136-018-1939-8. Epub 2018 Jul 20. PMID 30030674
- [Background] Aandstad A, Hageberg R, Holme IM, Anderssen SA. Objectively Measured Physical Activity in Home Guard Soldiers During Military Service and Civilian Life. Mil Med. 2016 Jul;181(7):693-700. doi: 10.7205/MILMED-D-15-00147. PMID 27391624
- [Background] Wynd CA, Bonnefil C, Harris JS. A comparison of health needs and personal health goals of Army Reserve Military and civilian employees. Mil Med. 2001 Jan;166(1):14-20. PMID 11197090
- [Background] Wynd CA, Ryan-Wenger NA. Factors predicting health behaviors among Army Reserve, active duty Army, and civilian hospital employees. Mil Med. 2004 Dec;169(12):942-7. doi: 10.7205/milmed.169.12.942. PMID 15646182
- [Background] Ballweg JA, Li L. Comparison of health habits of military personnel with civilian populations. Public Health Rep. 1989 Sep-Oct;104(5):498-509. PMID 2508180
- [Background] van Poppel MN, Chinapaw MJ, Mokkink LB, van Mechelen W, Terwee CB. Physical activity questionnaires for adults: a systematic review of measurement properties. Sports Med. 2010 Jul 1;40(7):565-600. doi: 10.2165/11531930-000000000-00000. PMID 20545381
- [Background] Peel C, Sawyer Baker P, Roth DL, Brown CJ, Brodner EV, Allman RM. Assessing mobility in older adults: the UAB Study of Aging Life-Space Assessment. Phys Ther. 2005 Oct;85(10):1008-119. PMID 16180950
- [Derived] Lee JW, Antonellis P, Fino PC, Peterka RJ, Wilhelm JL, Scanlan KT, Stojak ME, Brodsky JL, Monoli C, Weston AR, Liu W, Campbell KR, Schiltz K, Robinson I, Geisler CM, Chen S, Weightman MM, Hoppes CW, Dibble L, Chesnutt JC, King LA. Wearable technology to characterize and treat mild traumatic brain injury subtypes: Study protocol for a randomized controlled trial on biofeedback-based precision rehabilitation (SuBTyPE). PLoS One. 2026 Jan 30;21(1):e0340867. doi: 10.1371/journal.pone.0340867. eCollection 2026. PMID 41615970

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT06381674/Prot_SAP_ICF_004.pdf
  • Statistical Analysis Plan: Updated Statistical Analysis Document (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT06381674/SAP_003.pdf